CLINICAL TRIAL: NCT05518032
Title: A Phase 2 Study of Intravenous Pembrolizumab and Intratumorally Injected Autologous Dendritic Cells (DCs) in Refractory Colorectal Cancer (CRC)
Brief Title: Pembrolizumab and Autologous Dendritic Cells for the Treatment of Refractory Colorectal Cancer (CRC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: prioritization of studies
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I - 1670021; NCI-2022-04955 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I - 1670021 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Microsatellite Stable Colorectal Carcinoma; Recurrent Colorectal Carcinoma; Stage III Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Unresectable Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Biopsy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (pembrolizumab, autologous dendritic cells) (Experimental): Patients receive pembrolizumab IV on days 8, 29, 50, and 71, and autologous dendritic cells intratumorally on days 1 and 8 in the absence of disease progression or unacceptable toxicity. Patients may also receive an autologous dendritic cells intratumorally on day 50.
  Interventions: Procedure: Biopsy; Biological: Pembrolizumab; Biological: Therapeutic Autologous Dendritic Cells

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Therapeutic Autologous Dendritic Cells — Given intratumorally

SUMMARY:
The phase II trial tests whether pembrolizumab and dendritic cell-based treatment works to shrink tumors in patients with colorectal cancer that does not respond to treatment (refractory). Pembrolizumab, also referred to as an immune checkpoint inhibitor drug, works by targeting molecules that act as a check and balance system for immune responses. Immune checkpoint inhibitor drugs are designed to either "unleash" or "enhance" the cancer immune responses that already exist by either (1) blocking inhibitory molecules or by (2) activating stimulatory molecules. Dendritic cell-based treatment works by boosting the immune system (a system in our bodies that protects us against infection) to recognize and destroy the cancer cells. This investigational treatment targets cancer cells and is made from the patient's own blood cells. Giving pembrolizumab and dendritic cell-based treatment may help shrink tumors in patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the clinical efficacy of pembrolizumab in combination with intratumorally injected autologous dendritic cells (DCs) in refractory metastatic colorectal cancer (CRC).

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of pembrolizumab in combination with intratumorally injected autologous dendritic cells (DCs) in CRC patients.

II. To assess progression-free survival (PFS) in CRC patients receiving pembrolizumab in combination with intratumorally injected autologous dendritic cells (DCs).

III. To assess overall survival (OS) in CRC patients receiving pembrolizumab in combination with intratumorally injected autologous dendritic cells (DCs).

IV. To assess objective response as determined by Immune-related Response Evaluation Criteria in Solid Tumors (iRECIST).

EXPLORATORY OBJECTIVES:

I. To conduct correlative science studies including:

Ia. Comparison of the metastatic tissue specimen with regard to total numbers of infiltrating T cells, their CD4/CD8 ratios, frequencies of Tregs, and their expression of chemokine receptors.

Ib. Evaluate the local expression of T eff-attracting chemokines and T reg-favoring chemokines using immunofluorescence (IF) and reverse transcription-polymerase chain reaction (RT-PCR).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) on days 8, 29, 50, and 71, and autologous dendritic cells intratumorally on days 1 and 8 in the absence of disease progression or unacceptable toxicity. Patients may also receive an autologous dendritic cells intratumorally on day 50.

After completion study treatment, patients are followed up at 30 and 90 days, and then every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Recurrent and/or metastatic unresectable microsatellite stable (MSS) colorectal cancer
* At least 2 target lesions present per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 at least one of which is amenable to biopsy and injection
* Prior treatment with, contra-indication to, or refusal of a fluoropyrimidine, irinotecan, oxaliplatin and an anti-EGFR targeted therapy (if RAS wt), as well as avastin/bevacizumab
* PD-1/PD-L1/PD-L2 treatment naïve patients are eligible
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Platelet >= 75,000/uL
* Hemoglobin >= 8 g/dL (without transfusion in the past 14 days)
* Absolute neutrophil count (ANC) >= 1500/uL
* Estimated creatinine clearance (Cockcroft Gault) >= 30 mL/min/ for participant with creatinine levels > 1.5 x institutional upper limit of normal (ULN)
* Total bilirubin: =< 2 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 2 x ULN
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) =< 3 x institutional ULN (=< 5 x ULN for participants with liver metastases)
* Women of childbearing potential must agree to use acceptable birth control methods for the duration of the study and until persistence of the study drug is no longer detected in the peripheral blood: This may be a period of several years. Methods for acceptable birth control include condoms, diaphragm or cervical cap with spermicide, intrauterine device, and hormonal contraception; it is recommended that a combination of two methods be used

  * NOTE: If the risk of conception exists, patients must continue to use highly effective contraception for at least two years following the last study treatment administration
* A male participant must agree to use a contraception during the treatment period and for at least 1 year after the last dose of study treatment and refrain from donating sperm during this period
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients currently treated with systemic immunosuppressive agents. If a patient is currently on steroids, they must be on a steroid dose less than or equal to an equivalent prednisone dose of 10 mg daily
* Patients with active autoimmune disease, requiring ongoing immunosuppressive therapy or history of transplantation
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Has received prior chemotherapy or radiotherapy within 2 weeks of start of study intervention. All chemotherapy or radiation-related toxicities must be resolved to =< grade 1, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-CNS disease
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection. Note: No HIV testing is required
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected) infection. Note: no testing for hepatitis B and hepatitis C is required
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At 12 weeks
  Determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be estimated using a 90% confidence interval obtained by Jeffrey's prior method.

SECONDARY OUTCOMES:
Incidence of toxicities and adverse events | Up to 90 days after last dose
  Assessed as per Common Terminology Criteria for Adverse Events version 5.0 and tabulated by type and grade.
Progression-free survival | From initiation of study treatment regimen to disease progression or death from any cause, assessed up to 1 year
  Will be summarized using standard Kaplan-Meier methods, where estimates of median survival will be obtained with 90% confidence intervals.
Overall survival | From the time of treatment initiation until death from any cause, assessed up to 1 year
  Will be summarized using standard Kaplan-Meier methods, where estimates of median survival will be obtained with 90% confidence intervals.
Objective response rate | Up to 1 year
  Determined by Immune-related RECIST. Will be estimated using a 90% confidence interval obtained by Jeffrey's prior method.

CONTACTS AND LOCATIONS:
Overall Officials: Sarbajit Mukherjee, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States